CLINICAL TRIAL: NCT04186546
Title: Zephyr Valve Registry
Brief Title: Zephyr Valve Registry (ZEVR)
Acronym: ZEVR
Status: Active, not recruiting | Type: Observational
Sponsor: Pulmonx Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 630-0024-01
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Emphysema
Keywords: emphysema; endobronchial valve; treatments; pulmonary rehabilitation; lung volume reduction
MeSH Terms: conditions — Emphysema | interventions — Pneumonectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Cases: Zephyr Valve Procedure
  Interventions: Device: Zephyr Valve Procedure

INTERVENTIONS:
Device: Zephyr Valve Procedure — The Pulmonx Zephyr Endobronchial Valve is an implantable bronchial valve intended to decrease volume in targeted regions of the lung. It is indicated for the treatment of patients with severe emphysema. The Zephyr Valves are placed in the diseased region of the lung using bronchoscopy. As the diseased region of the lung shrinks in size, healthier regions may expand and function more efficiently, resulting in improved breathing.
  Other Names: Zephyr Endobronchial Valve; Endobronchial Valve; Bronchoscopic Lung Volume Reduction; BLVR

SUMMARY:
The purpose of this Post-Approval Registry is to gather ongoing safety and effectiveness assessment of the Zephyr Valve treatment in a real-world setting.

DETAILED DESCRIPTION:
The Zephyr Valve Registry (ZEVR) is a multi-center, single-arm, prospective Registry. The objective of this Registry is to provide ongoing safety and effectiveness assessment of the Zephyr Valve treatment of patients with hyperinflation associated with severe emphysema, in regions of the lung that have little to no collateral ventilation.

Approximately 150 patients undergoing Zephyr Valve treatment in the commercial setting will be enrolled and followed out to 3 years. Assessments will be conducted at 45-days, 6-months, 12-months, 24-months and 36-months post-procedure. The Zephyr Valve Registry will be conducted at a minimum of 5, and a maximum of 10 clinical sites.

Subjects prescribed Zephyr Valve treatment for their emphysema will be consented and will be enrolled only after determination of little to no collateral ventilation between target and ipsilateral lobes. Safety and effectiveness of the Zephyr Valve treatment will be evaluated post-treatment based on data collected out to 3 years after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with severe emphysema considered appropriate for the procedure by the physician.
* Subjects who signed an Informed Consent Form to allow data collection.

Exclusion Criteria:

• Subjects determined to have collateral ventilation between the target(s) and ipsilateral lobe(s).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Registry population will be comprised of subjects with hyperinflation of the lungs due to severe emphysema that are prescribed the Zephyr Valve treatment by their physician and confirmed to have little to no collateral ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence Rate of Pneumothorax from Baseline to 45-days post-procedure | Baseline to 45-days post-procedure
  The percentage of study participants undergoing the Zephyr Valve Procedure who develop a pneumothorax from the date of the procedure to 45-day post intervention.
Incidence Rate of Serious Adverse Events (SAEs) of Interest from Baseline to 3 years post-procedure | Baseline to 3 years post-procedure
  The percentage of study participants who experience a device and/or procedure related SAE including but not limited chronic obstructive pulmonary disease (COPD) exacerbation, hemoptysis, pneumonia, respiratory failure, Valve expectoration and Valve migration

SECONDARY OUTCOMES:
Absolute Change in Treated Lobar Volume Reduction (TLVR) after 45-days post-procedure | At baseline and after 45-days post-procedure
  The Treated Lobe Volume Reduction (TLVR) will be evaluated by quantitative analysis of high-resolution computed tomography (HRCT) scans at Baseline and at 45-days post-valve placement to measure the treated lobe volume reduction.
Percent Change in Treated Lobar Volume Reduction (TLVR) after 45-days post-procedure | At baseline and after 45-days post-procedure
  The Treated Lobe Volume Reduction (TLVR) will be evaluated by quantitative analysis of HRCT scans at Baseline and at 45-days post-valve placement to measure the treated lobe volume reduction.
Absolute Change in Forced Expiratory Volume in 1 second FEV1 (L) Post Bronchodilator from baseline to 6-months, 12-months, 24-months and 36-months post-procedure | At baseline, 6-months, 12-months, 24-months and 36-months post-procedure
  The mean absolute change in FEV1(L) relative to Baseline at 6-months, 12-months, 24-months and 36-months post procedure
Percent Change in Forced Expiratory Volume in 1 second FEV1 (L) Post Bronchodilator from baseline to 6-months, 12-months, 24-months and 36-months post-procedure | At baseline, 6-months, 12-months, 24-months and 36-months post-procedure
  The mean percent change in FEV1(L) relative to Baseline at 6-months, 12-months, 24-months and 36-months post procedure
Absolute Change in Forced Expiratory Volume in 1 second FEV1 (% Predicted) Post Bronchodilator from baseline to 6-months, 12-months, 24-months and 36-months post-procedure | At baseline, 6-months, 12-months, 24-months and 36-months post-procedure
  The mean absolute change in FEV1(% Predicted) relative to Baseline at 6-months, 12-months, 24-months and 36-months post procedure.
Percent Change in Forced Expiratory Volume in 1 second FEV1 (% Predicted) Post Bronchodilator from baseline to 6-months, 12-months, 24-months and 36-months post-procedure | At baseline, 6-months, 12-months, 24-months and 36-months post-procedure
  Mean percent change in FEV1(% Predicted) relative to Baseline at 6-months, 12-months, 24-months and 36-months post-procedure
Absolute Change in Six-Minute Walk Distance (6MWD) from baseline to 6-months and 12-months post-procedure | At baseline, 6-months and 12-months
  Mean absolute change in the 6MWD from Baseline to 6-months and 12-months post-procedure.
Percent Change in Six-Minute Walk Distance (6MWD) from baseline to 6-months and 12-months post-procedure | At baseline, 6-months and 12-months
  Mean percent change in the 6MWD from Baseline to 6-months and 12-months post-procedure.
Absolute Change in St. George's Respiratory Questionnaire (SGRQ) Total Score from baseline to 6-months and 12-months post-procedure | At baseline, 6-months and 12-months
  Mean absolute change in the St. George's Respiratory Questionnaire Total Score from Baseline to 6-months and 12-months post-procedure. Scores range from 0 to 100, with higher scores indicating more limitations.
Percent Change in St. George's Respiratory Questionnaire (SGRQ) Total Score from baseline to 6-months and 12-months post-procedure | At baseline, 6-months and 12-months
  Mean percent change in the St. George's Respiratory Questionnaire Total Score from Baseline to 6-months and 12-months post-procedure. Scores range from 0 to 100, with higher scores indicating more limitations.
Absolute Change in BODE Index Total Score from baseline to 6-months and 12-months post-procedure | At baseline, 6-months and 12-months
  BODE stands for Body mass index, airflow Obstruction, Dyspnea and Exercise capacity. The BODE Index is a tool used to predict the death risk by using an algorithm that considers the following variables: body mass index (BMI, B), airflow obstruction (O) as measured by the post-bronchodilator FEV1 (percentage of predicted value), dyspnea (D) assessed by the modified Medical Research Council (MMRC) score, and exercise tolerance (E) measured by 6 minute walking distance. These variables are graded 0 to 3 (0 or 1 for BMI) and summed to give a total score between 0 and 10. The resulting score is called the BODE index, with higher scores indicating a greater risk of death. The mean absolute change in the BODE score will be calculated from baseline scores compared to the BODE score at 6 months and 12 months post procedure.
Percent change in BODE Index Total Score from baseline to 6-months and 12-months post-procedure | At baseline, 6-months and 12-months
  BODE stands for Body mass index, airflow Obstruction, Dyspnea and Exercise capacity. The BODE Index is a tool used to predict the death risk by using an algorithm that considers the following variables: body mass index (BMI, B), airflow obstruction (O) as measured by the post-bronchodilator FEV1 (percentage of predicted value), dyspnea (D) assessed by the modified Medical Research Council (MMRC) score, and exercise tolerance (E) measured by 6 minute walking distance. These variables are graded 0 to 3 (0 or 1 for BMI) and summed to give a total score between 0 and 10. The resulting score is called the BODE index, with higher scores indicating a greater risk of death. The mean percent change in the BODE score will be calculated from baseline scores compared to the BODE score at 6 months and 12 months post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Kutzavitch, PhD, Study Director — Pulmonx Corporation
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Chicago, Chicago, Illinois
  - Northwestern Medicine, Winfield, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - The Lung Center, DuBois, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Houston Methodist, Houston, Texas
  - Inova Health, Fairfax, Virginia
  - Froedtert Memorial-Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Valipour A, Slebos DJ, Herth F, Darwiche K, Wagner M, Ficker JH, Petermann C, Hubner RH, Stanzel F, Eberhardt R; IMPACT Study Team. Endobronchial Valve Therapy in Patients with Homogeneous Emphysema. Results from the IMPACT Study. Am J Respir Crit Care Med. 2016 Nov 1;194(9):1073-1082. doi: 10.1164/rccm.201607-1383OC. PMID 27580428
- [Background] Klooster K, ten Hacken NH, Hartman JE, Kerstjens HA, van Rikxoort EM, Slebos DJ. Endobronchial Valves for Emphysema without Interlobar Collateral Ventilation. N Engl J Med. 2015 Dec 10;373(24):2325-35. doi: 10.1056/NEJMoa1507807. PMID 26650153
- [Background] Klooster K, Hartman JE, Ten Hacken NH, Slebos DJ. One-Year Follow-Up after Endobronchial Valve Treatment in Patients with Emphysema without Collateral Ventilation Treated in the STELVIO Trial. Respiration. 2017;93(2):112-121. doi: 10.1159/000453529. Epub 2016 Dec 15. PMID 27974713
- [Background] Hartman JE, Klooster K, Slebos DJ, Ten Hacken NH. Improvement of physical activity after endobronchial valve treatment in emphysema patients. Respir Med. 2016 Aug;117:116-21. doi: 10.1016/j.rmed.2016.06.009. Epub 2016 Jun 9. PMID 27492521
- [Background] Davey C, Zoumot Z, Jordan S, McNulty WH, Carr DH, Hind MD, Hansell DM, Rubens MB, Banya W, Polkey MI, Shah PL, Hopkinson NS. Bronchoscopic lung volume reduction with endobronchial valves for patients with heterogeneous emphysema and intact interlobar fissures (the BeLieVeR-HIFi study): a randomised controlled trial. Lancet. 2015 Sep 12;386(9998):1066-73. doi: 10.1016/S0140-6736(15)60001-0. Epub 2015 Jun 23. PMID 26116485
- [Background] Zoumot Z, Davey C, Jordan S, McNulty WH, Carr DH, Hind MD, Polkey MI, Shah PL, Hopkinson NS. Endobronchial valves for patients with heterogeneous emphysema and without interlobar collateral ventilation: open label treatment following the BeLieVeR-HIFi study. Thorax. 2017 Mar;72(3):277-279. doi: 10.1136/thoraxjnl-2016-208865. Epub 2016 Dec 20. PMID 27999170
- [Background] Sciurba FC, Ernst A, Herth FJ, Strange C, Criner GJ, Marquette CH, Kovitz KL, Chiacchierini RP, Goldin J, McLennan G; VENT Study Research Group. A randomized study of endobronchial valves for advanced emphysema. N Engl J Med. 2010 Sep 23;363(13):1233-44. doi: 10.1056/NEJMoa0900928. PMID 20860505
- [Background] Herth FJ, Noppen M, Valipour A, Leroy S, Vergnon JM, Ficker JH, Egan JJ, Gasparini S, Agusti C, Holmes-Higgin D, Ernst A; International VENT Study Group. Efficacy predictors of lung volume reduction with Zephyr valves in a European cohort. Eur Respir J. 2012 Jun;39(6):1334-42. doi: 10.1183/09031936.00161611. Epub 2012 Jan 26. PMID 22282552
- [Background] Skowasch D, Fertl A, Schwick B, Schafer H, Hellmann A, Herth FJ; LIVE Study Investigators. A Long-Term Follow-Up Investigation of Endobronchial Valves in Emphysema (the LIVE Study): Study Protocol and Six-Month Interim Analysis Results of a Prospective Five-Year Observational Study. Respiration. 2016;92(2):118-26. doi: 10.1159/000448119. Epub 2016 Aug 24. PMID 27562904
- [Background] Criner GJ, Sue R, Wright S, Dransfield M, Rivas-Perez H, Wiese T, Sciurba FC, Shah PL, Wahidi MM, de Oliveira HG, Morrissey B, Cardoso PFG, Hays S, Majid A, Pastis N Jr, Kopas L, Vollenweider M, McFadden PM, Machuzak M, Hsia DW, Sung A, Jarad N, Kornaszewska M, Hazelrigg S, Krishna G, Armstrong B, Shargill NS, Slebos DJ; LIBERATE Study Group. A Multicenter Randomized Controlled Trial of Zephyr Endobronchial Valve Treatment in Heterogeneous Emphysema (LIBERATE). Am J Respir Crit Care Med. 2018 Nov 1;198(9):1151-1164. doi: 10.1164/rccm.201803-0590OC. PMID 29787288
- [Background] Kemp SV, Slebos DJ, Kirk A, Kornaszewska M, Carron K, Ek L, Broman G, Hillerdal G, Mal H, Pison C, Briault A, Downer N, Darwiche K, Rao J, Hubner RH, Ruwwe-Glosenkamp C, Trosini-Desert V, Eberhardt R, Herth FJ, Derom E, Malfait T, Shah PL, Garner JL, Ten Hacken NH, Fallouh H, Leroy S, Marquette CH; TRANSFORM Study Team *. A Multicenter Randomized Controlled Trial of Zephyr Endobronchial Valve Treatment in Heterogeneous Emphysema (TRANSFORM). Am J Respir Crit Care Med. 2017 Dec 15;196(12):1535-1543. doi: 10.1164/rccm.201707-1327OC. PMID 28885054